CLINICAL TRIAL: NCT05161767
Title: Shifting Away From Pain: Neurocognitive Approach to Explain and Predict Recovery Following Whiplash Injury
Status: Terminated | Type: Observational
Why Stopped: Difficult recruitment of acute patients via emergency services due to COVID-19. The required sample size was consequently not reached within the PhD period of the involved researchers.
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: B670201941074
Record Dates: First submitted 2021-12-03; First posted 2021-12-17 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Whiplash Injuries
Keywords: whiplash; chronic pain; neuroimaging
MeSH Terms: conditions — Whiplash Injuries; Chronic Pain | interventions — Neuroimaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Recovered group: This will group will consists of people who have a remission of their symptoms at 6-months follow-up after whiplash injury.
  Interventions: Diagnostic Test: Brain MRI (neuroimaging)
- non-recovered group: This will group will consists of people who develop persistent symptoms at 6-months follow-up after whiplash injury.
  Interventions: Diagnostic Test: Brain MRI (neuroimaging)

INTERVENTIONS:
Diagnostic Test: Brain MRI (neuroimaging) — Structural and functional brain scans will be taken.

SUMMARY:
Around half of the patients with neck pain after trauma (whiplash) will develop chronic pain. Understanding the transition from acute to chronic pain after whiplash is a priority since will help to identify those which patients are likely to fully recover and who do not. In the last years, there have been a call for an investigation of new biomarkers; particularly in brain structure and function. Alterations in the structure of the brain (gray matter, white matter and cortical thickness) as well as the brain function have been found in people with chronic WAD; which are also correlated with pain, disability and symptoms of central sensitization such as hyperalgesia. Previous research has found structural and functional brain differences between people who develop chronic low back pain compared to those who recovered; but research in this vein is still lacking in people with whiplash. Consequently, this study aims to examine the neural correlates of recovery following whiplash injury.

DETAILED DESCRIPTION:
This study aims to investigate whether or not there are differences in brain structure and function between people who recover after whiplash and those who do not. Thus, patients with acute neck pain after whiplash will be recruited. Also, a pain-free age- and sex-matched control group will be recruited for comparison.

A longitudinal prospective study will be conducted with two follow-up measurements (3 and 6 months). All measurements will take place at University Hospital of Ghent (UZ Gent), Ghent (Belgium). MRI measures will be taken at baseline (<4 weeks after the accident) and 6-months follow-up. The 3-months follow-up will only consist of the assessment of the online questionnaires; so, patients will not be required to come to UZ Gent.

ELIGIBILITY:
Whiplash patients

Inclusion Criteria:

* Neck pain within 4 weeks after the trauma
* Native Dutch speaker
* Refraining from consuming caffeine, alcohol and nicotine in the hour before the MRI scans in both measurement times

Exclusion Criteria:

* Neuropathic pain
* Being pregnant
* A history of a chronic pain syndrome
* Chronic fatigue syndrome
* Fibromyalgia
* Cardiovascular disorders
* Epilepsy
* Endocrinological disorders
* Rheumatic disorders
* Psychiatric disorders
* History of neck surgery
* Loss of consciousness during/after the whiplash trauma
* MRI incompatible health condition (e.g., pacemaker, metal prosthetic devices)
* Claustrophobia.

Healthy volunteers: (matched for age and gender). Additional exclusion criteria include for healthy volunteers

* a history of a chronic pain syndrome
* a pain condition in the last six months for which treatment was sought

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Whiplash injury is a type of neck injury caused by sudden movement of the head forwards, backwards or sideways (i.e. motor vehicle accident)
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Blood oxygenation level dependent (BOLD) signal (functional MRI) during picture imagination task and during resting state | Baseline and 6-months follow-up
  Change between baseline assessment (within 4 weeks after the trauma) and the 6-months follow-up assessment.
Structural MRI measures (i.e., grey and white matter) | Baseline and 6-months follow-up
  Change between baseline assessment (within 4 weeks after the trauma) and the 6-months follow-up assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Iris Coppieters, PhD, Principal Investigator — Vrije Universiteit Brussel, KU Leuven
Locations (1):
- Department of rehabilitation sciences (Ghent University), Ghent, Belgium